CLINICAL TRIAL: NCT05291052
Title: A Single-arm, Open-label Clinical Study of Combined Therapy of Tisleizumab , Lenvatinib and XELOX Regimen (Oxaliplatin Combined With Capecitabine) in the First-line Treatment of Advanced and Unresectable Biliary Tract Tumors
Brief Title: Tisleizumab Combined With Lenvatinib and XELOX Regimen (Oxaliplatin Combined With Capecitabine) in the First-line Treatment of Advanced and Unresectable Biliary Tract Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tis-BTC-001
Record Dates: First submitted 2022-03-14; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Biliary Tract Tumor
MeSH Terms: interventions — tislelizumab; lenvatinib; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIS combined therapy (Experimental): All patients will be treated with the combination of tisleizumab , lenvatinib and XELOX regimen (oxaliplatin combined with capecitabine) until disease progression , unacceptable toxicity, death or the patient meets any other discontinuation criteria described in the protocol, whichever occurs first. Subjects can receive up to 8 cycles of the XELOX regimen. For subjects who are intolerant to XELOX regimen or have stable disease or objective response after complete 8 cycles of XELOX regimen, treatment with tisleizumab and lenvatinib will be continued until tumor progression or for a maximum of 2 years.
  Interventions: Drug: Tislelizumab; Drug: Lenvatinib; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Tislelizumab — Tisleizumab 200 mg intravenously (IV) every 3 weeks (Q3W) ,D1
Drug: Lenvatinib — Lenvatinib 8 mg (for patient weight < 60 kg) or 12 mg (for patient weight ≥ 60 kg), orally, QD, D1-21, Q3W
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2, IV， D1，Q3W
  Subjects can receive up to 8 cycles of the XELOX regimen (Oxaliplatin and Capecitabine). For subjects who are intolerant to XELOX regimen or have stable disease or objective response after complete 8 cycles of XELOX regimen, treatment with tisleizumab and lenvatinib will be continued until tumor progression or for a maximum of 2 years.
Drug: Capecitabine — Capecitabine 1000 mg/m2, orally, BID, D1-14, Q3W
  Subjects can receive up to 8 cycles of the XELOX regimen (Oxaliplatin and Capecitabine). For subjects who are intolerant to XELOX regimen or have stable disease or objective response after complete 8 cycles of XELOX regimen, treatment with tisleizumab and lenvatinib will be continued until tumor progression or for a maximum of 2 years.

SUMMARY:
This study is a single-center, single-arm, open-label clinical study. All patients with advanced and unresectable biliary tract tumors will be treated with the combination of tisleizumab, lenvatinib and XELOX regimen (oxaliplatin plus capecitabine) until disease progression , unacceptable toxicity, death or the patient meets any other discontinuation criteria described in the protocol, whichever occurs first. Subjects can receive up to 8 cycles of the XELOX regimen. For subjects who are intolerant to XELOX regimen or have stable disease or objective response after complete 8 cycles of XELOX regimen, treatment with tisleizumab and lenvatinib will be continued until tumor progression or for a maximum of 2 years. Patients will be closely monitored for safety and tolerability throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, a patient must meet all of the following criteria:

  1. Able to provide written informed consent and able to understand and agree to comply with study requirements and assessment schedules
  2. Histologically or cytologically confirmed unresectable or postoperative recurrent locally advanced or metastatic biliary tract tumors, including cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer;
  3. Aged 18-75 years old, male or female;
  4. Eastern Cooperative Oncology Group (ECOG) fitness status score (PS score) 0-1;
  5. Expected survival ≥ 3 months;
  6. At least one measurable lesion according to RECIST V1.1;
  7. No previous systemic therapy, including chemotherapy, targeted therapy, immunotherapy;
  8. Adequate organ function as indicated by the following laboratory values ≤ 7 days prior to the first dose of study drug:

     a. Patients must not have required a transfusion of blood product or growth factor support within the 14 days before sample collection during the Screening Period and met all of the following criteria:

     i. Absolute neutrophil count（ANC）≥ 1.5 × 10^9/L

     ii. Platelets ≥ 75 × 10^9/L

     iii. Hemoglobin ≥ 90 g/L

     b. Serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance > 50 μmol/L

     c. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 × ULN; if there is a lesion in liver, ALT or AST ≤ 5 × ULN;

     d. Serum total bilirubin ≤ 1.5 × ULN;

     e. International normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 × ULN

     f. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN

     g. Cardiac Doppler ultrasound evaluation score (LVEF) ≥ 50%.
  9. Patients with positive hepatitis B surface antigen (HBsAg) or previous history of HBV infection must receive antiviral agents before the first dose of study drug and continue treatment during the study.
  10. Females of childbearing potential must agree to practice highly effective contraception during the study and for ≥ 120 days after the last dose of study drug and have a negative serum pregnancy test ≤ 7 days of the first study drug administration
  11. Nonsterilized male patients must agree to practice highly effective contraception for the duration of the study and for ≥ 120 days after study drug administration
  12. Good compliance and family agrees to cooperate with survival follow-up.

Exclusion Criteria:

* To be eligible to participate in this study, a patient cannot meet any of the following exclusion criteria:

  1. Any active malignancy ≤ 2 years prior to the first dose of study drug, except the specific cancers evaluated in this study and any curatively treated locally recurrent cancer (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast).
  2. Participation in other clinical trials within four weeks prior to the first dose of study drug;
  3. Patients with any evidence or history of bleeding diatheses regardless of severity; patients with any bleeding or bleeding event ≥ CTCAE grade 3 within 4 weeks before the first dose; patients with gastrointestinal diseases such as unhealed wound, fracture, active gastric and duodenal ulcer, ulcerative colitis or active bleeding of unresected tumor, or other conditions that may cause gastrointestinal bleeding and perforation judged by the investigator;
  4. Patients with uncontrolled brain metastasis, spinal cord compression, carcinomatous meningitis or brain or leptomeningeal disease found by CT or MRI within 4 weeks before the first dose of study drug;
  5. Patients with any severe and/or uncontrolled disease, including: a) patients with unsatisfactory blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg); b) unstable angina pectoris, myocardial infarction, ≥ grade 2 congestive heart failure, or arrhythmia requiring treatment (including QTc ≥ 480 ms) within 6 months before the first dose of study drug; c) severe chronic or active infection (including tuberculosis infection, etc.) requiring systemic antibacterial, antifungal or antiviral therapy within 14 days before the first dose of study drug, Note: patients with viral hepatitis are allowed to receive antiviral therapy; d) positive HIV test; e) poor control of diabetes (fasting blood glucose ≥ CTCAE grade 2); f) urine routine indicating urine protein ≥ 1 +, and confirmed 24-hour urine protein quantification > 1.0 g;
  6. Patients with any active autoimmune disease or a history of autoimmune disease (such as, but not limited: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; patients with asthma requiring medical intervention with bronchodilators can not be included); patients with the following are allowed: vitiligo, psoriasis, alopecia without systemic treatment, well-controlled type I diabetes, hypothyroidism after replacement therapy;
  7. If HCV RNA is detectable, the presence of HCV infection is confirmed and such patients are not eligible;
  8. Uncontrolled pleural effusion, pericardial effusion or peritoneal effusion requiring frequent drainage or medical intervention (clinically significant recurrence,requiring additional intervention within two weeks after intervention, excluding exfoliative cytology of exudates) within 7 days before the first dose of study drug;
  9. Has any condition that required systemic treatment with corticosteroids (> 10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days before the first dose of study drug.
  10. Use of Chinese herbal medicines or Chinese patent medicines with antitumor activity approved by the China National Medical Products Administration (NMPA), regardless of the type of cancer, within 14 days before the first dose of study drug
  11. Has been administered a live vaccine within 28 days prior to study drug administration
  12. Has a History of severe hypersensitivity reaction or any contraindication to any component of the tislelizumab or lenvatinib formulation or any component of the container;
  13. Patients with concomitant diseases that seriously jeopardize the patient's safety or affect the patient's completion of the study judged by the investigator;
  14. Pregnant and lactating women;
  15. Malabsorption syndrome or inability to take oral medications for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) per RECIST v1.1 assessed by investigator | 12months
  It is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR.
Safety as measured by the rate of AEs | 12months
  Safety will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

SECONDARY OUTCOMES:
ORR per iRECIST by the investigator | 12months
  ORR assessed by the investigator according to iRECIST
Disease control rate (DCR) | 12months
  Disease control rate (DCR) assessed by the investigator according to RECIST v1.1 and iRECIST
duration of response (DOR) | 12months
  DOR assessed by the investigator according to RECIST v1.1 and iRECIST
progression-free survival (PFS) | 12months
  progression-free survival (PFS) assessed by the investigator according to RECIST v1.1 and iRECIST
Overall survival (OS) | 24months
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China